CLINICAL TRIAL: NCT02971592
Title: Estimation of Therapeutic Effect of MDcure on Patients With Chronic Back Pain
Brief Title: Estimation of Therapeutic Effect of MDcure on Patients With Chronic Lower Back Pain
Acronym: E_MDcure_LBP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assuta Medical Center (Other)
Collaborators: Aerotel Ltd (Industry)
Responsible Party: Principal Investigator, Dr. Eran Segal, Principal Investigator, Assuta Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0047-16-ASM
Record Dates: First submitted 2016-11-20; First posted 2016-11-23 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Back Pain Lower Back Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Device: MDcure
- Placebo (Placebo Comparator)
  Interventions: Other: Mock Device

INTERVENTIONS:
Device: MDcure — reception of real working MDcure - device that does apply the electromagnetic field
  Arms: Experimental
Other: Mock Device — reception of device that does not apply the electromagnetic field
  Arms: Placebo

SUMMARY:
This study will assess the therapeutic effect of MDcure® device. MDcure® is an FDA Class 1 listed medical device, produced to ISO-13485 standards, that delivers extremely low intensity (nano Tesla; 10-9) and low frequencies (1-100 Hertz) electromagnetic fields (EMF) intended to reduce muscular aches and pains particularly of the lower back.

assessing the reduction of lower back pain. Half of participants will receive the MDcure device, while the other half will receive a mock device.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-75
* Patients with chronic lower back for more then 3 month
* Patients who scored over 21% and below 60% in the Oswestry questionnaire

Exclusion Criteria:

* A neurological deficient in lower limbs
* Patients who scored more than 60% on the Oswestry questionnaire.
* Patients who underwent surgical intervention in spine including metal implant in lower back
* Patients diagnosed with cancer
* Patients with any type of vertebral fracture
* Patients who received steroid injection less then a month prior to starting the experiment
* Patients treated with steroids as a preventive treatment on a regular basis
* Patients using narcotic drugs for over a six month period or cannabis or any other sort of narcotic drug for over a six month period prior to their enrollment in the study
* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Improvement in pain in experiment group | 6 weeks
  Assessment of rate of patients from the experiment group who report improvement in pain above 20% in Oswestry scale
Improvement in pain in placebo group | 6 weeks
  Assessment of rate of patients from the placebo group who report improvement in pain above 20% in Oswestry scale

SECONDARY OUTCOMES:
Assess period of time to attain improvement | maximum of 6 weeks
  Assess the duration period of improvement, starting from the beginning of the experiment up to the point where 20% improvement is attained

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta Medical Centers - Ramat Hahyal, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No